CLINICAL TRIAL: NCT03344653
Title: Onyx ONE Study; A Randomized Controlled Trial With Resolute Onyx in One Month Dual Antiplatelet Therapy (DAPT) for High-Bleeding Risk Patients
Brief Title: A Randomized Controlled Trial With Resolute Onyx in One Month Dual Antiplatelet Therapy (DAPT) for High-Bleeding Risk Patients
Acronym: Onyx ONE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Vascular (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MDT17054RES007
Record Dates: First submitted 2017-10-20; First posted 2017-11-17 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-12

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Prospective, multi-center, blinded, randomized, controlled study enrolling eligible subjects at global centers. The enrollment period is anticipated to be approximately 14 months.
Who Masked: Participant
Masking Description: Subjects will be randomized at a 1:1 ratio to treatment with Resolute Onyx stent or the BioFreedom stent (control).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Resolute Onyx stent (Active Comparator): Subjects who fulfill the inclusion criteria and none of the exclusion criteria will be randomly allocated in a 1:1 fashion to treatment with a Resolute Onyx stent or the BioFreedom stent followed by 1-month DAPT. Subjects implanted with the Resolute Onyx stent will be assessed for non-inferiority compared to those implanted with the BioFreedom stent using a composite safety endpoint of cardiac death, myocardial infarction, and definite/probable stent thrombosis, at 1 year post-procedure.
  Interventions: Device: Medtronic Resolute Onyx Zotarolimus-Eluting Coronary Stent System
- BioFreedom stent (Active Comparator): Subjects who fulfill the inclusion criteria and none of the exclusion criteria will be randomly allocated in a 1:1 fashion to treatment with a Resolute Onyx stent or the BioFreedom stent followed by 1-month DAPT. Subjects implanted with the Resolute Onyx stent will be assessed for non-inferiority compared to those implanted with the BioFreedom stent using a composite safety endpoint of cardiac death, myocardial infarction, and definite/probable stent thrombosis, at 1 year post-procedure.
  Interventions: Device: Biosensors BioFreedom BA9 Drug Coated Coronary Stent

INTERVENTIONS:
Device: Medtronic Resolute Onyx Zotarolimus-Eluting Coronary Stent System — Medtronic Resolute Onyx Zotarolimus-Eluting Coronary Stent System Treatment Followed by 1 month DAPT
  Arms: Resolute Onyx stent
Device: Biosensors BioFreedom BA9 Drug Coated Coronary Stent — Biosensors BioFreedom BA9 Drug Coated Coronary Stent Followed by 1 month DAPT
  Arms: BioFreedom stent

SUMMARY:
The purpose of this study is to evaluate the clinical safety and effectiveness of the Resolute Onyx stent in subjects deemed at high risk for bleeding and/or medically unsuitable for more than 1 month DAPT treatment receiving reduced duration (1 month) of DAPT following stent implantation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 75 years old
* Any prior documented intracerebral bleed
* Any documented stroke in the last 12 months
* Hospital admission for bleeding during the prior 12 months
* Non-skin cancer diagnosed or treated ≤3 years
* Planned surgery within the next 12 months
* Renal failure defined as: Creatinine clearance <40 ml/min
* Thrombocytopenia (PLT <100,000/mm3)
* Severe chronic liver disease defined as: subjects who have developed any of the following: variceal hemorrhage, ascites, hepatic encephalopathy or jaundice

Exclusion Criteria:

* Pregnant and breastfeeding women
* Subjects requiring a planned PCI procedure after 1 month of index procedure
* Active bleeding at the time of inclusion
* Cardiogenic shock
* A known hypersensitivity or contraindication to aspirin, heparin and bivalirudin, P2Y12 inhibitors, mTOR inhibiting drugs such as zotarolimus, Biolimus A9 (or its derivatives), cobalt, nickel, platinum, iridium, chromium, molybdenum, polymer coatings (eg, BioLinx™), stainless steel (or other metal ions found in 316L stainless steel), zinc, or a sensitivity to contrast media, which cannot be adequately pre-medicated.
* PCI during the previous 6 months for a lesion other than the target lesion of the index procedure
* Participation in another clinical study within 12 months after index procedure
* Subjects with life expectancy of less than 2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Actual)
Dates: Start 2017-11-02 (Actual); Primary Completion 2018-09-27 (Actual); Study Completion 2020-10-09 (Actual)

PRIMARY OUTCOMES:
Composite endpoint: Cardiac Death, Myocardial Infarction, or Stent Thrombosis | 1 year post-procedure
  Powered for non-inferiority against BioFreedom (control), is a composite of cardiac death, myocardial infarction and definite/probable stent thrombosis. The combined clinical outcome of cardiac death, MI or stent thrombosis

SECONDARY OUTCOMES:
Target Lesion Failure | 2 year post-procedure
  Defined as cardiac death, target vessel myocardial infarction (Q wave and non Q wave), or clinically driven target lesion revascularization(TLR) by percutaneous or surgical methods
Procedure Success | 2 year post-procedure
  Attainment of <30% residual stenosis by QCA (or <20% by visual assessment) AND TIMI flow 3 after the procedure, using any percutaneous method without the occurrence of MACE during the hospital stay.
Cardiac Death | 2 year post- procedure
  All deaths including cardiac death
Major Cardiac Event | 2 year post- procedure
  Major adverse cardiac event (MACE) defined as composite of death, myocardial infarction, or repeat target lesion revascularization (clinically driven) by percutaneous or surgical methods
Myocardial Infarction | 2 year post-procedure
  All myocardial infarction including Target Vessel Myocardial Infarction (TVMI)
Target Vessel Failure | 2 year post-procedure
  Target vessel failure (TVF) defined as composite of cardiac death, target vessel myocardial infarction, or clinically-driven target vessel revascularization (TVR) by percutaneous or surgical methods.
Revascularization | 2 year post-procedure
  All revascularizations (TLR, TVR and non-TVR)
Stent Thrombosis | 2 year post-procedure
  Stent thrombosis (per Academic Research Consortium (ARC) definition)
Bleeding | 2 year post-procedure
  Bleeding per BARC criteria
Stroke | 2 year post-procedure
  Stroke
Lesion Success | 2 year post-procedure
  The attainment of <30% residual stenosis by QCA (or < 20% by visual assessment) AND TIMI flow 3 after the procedure, using any percutaneous method
Device success | 2 year post-procedure
  Attainment of <30% residual stenosis by QCA (or <20% by visual assessment) AND TIMI flow 3 after the procedure, using the assigned device only.

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Windecker, MD, Principal Investigator — Bern University Hospital, Bern, Switzerland; Azeem Latib, MD, Principal Investigator — San Raffaele Scientific Institute, Milan, Italy; Elvin Kedhi, MD, Principal Investigator — Isala Zwolle, Netherlands
Locations (88):
- Australia (11):
  - Royal North Shore Hospital, Saint Leonards, New South Wales
  - Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - Bundaberg Cardiology - Friendly Society Private Hospital, Bundaberg, Queensland
  - Cairns Hospital, Cairns, Queensland
  - The Prince Charles Hospital, Chermside, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Adelaide Cardiology, Adelaide, South Australia
  - Flinders Medical Centre, Bedford Park, South Australia
  - Saint Vincent's Hospital (Melbourne), Fitzroy, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
- Austria (3):
  - LKH - Universitätsklinikum Graz, Graz
  - A.ö. Landeskrankenhaus - Universitätskliniken Innsbruck, Innsbruck
  - Allgemeines Krankenhaus - Universitätskliniken Wien, Vienna
- Belgium (3):
  - C.H.U. de Charleroi, Charleroi
  - UZ Leuven - Campus Gasthuisberg, Leuven
  - CHU de Liège - Hôpital du Sart Tilman, Liège
- Acibadem City Clinic, Sofia, Bulgaria
- France (2):
  - Clinique Axium, Aix-en-Provence
  - Hôpital Privé Jacques Cartier, Massy
- Hong Kong (2):
  - Queen Elizabeth Hospital (Hong Kong), Hong Kong
  - Queen Mary Hospital, Hong Kong
- Galway University Hospitals - University Hospital Galway (UHG), Galway, Ireland
- Italy (5):
  - Azienda Ospedaliera Bolognini Seriate - Ospedale Bolognini, Seriate, Bergamo
  - Presidio Ospedaliero Ferrarotto Alessi, Catania
  - San Raffaele Scientific Institute, Milan
  - Centro Cardiologico Monzino, Milan
  - Umberto I - Policlinico di Roma, Roma
- Latvia (2):
  - Paula Stradina Kliniska universitates slimnica, Riga
  - Riga East University Hospital, Riga
- Lithuania (2):
  - Hospital of Lithuanian University of Health Sciences Kauno Klinikos, Kaunas
  - Vilnius University Hospital Santariskiu Klinikos, Vilnius
- Malaysia (5):
  - Queen Elizabeth II Hospital, Kota Kinabalu, Sabah
  - Sarawak Heart Centre, Kuching, Sarawak
  - Hospital Serdang, Kajang, Selangor
  - Sarawak Heart Centre, Kota Kinabalu
  - Institut Jantung Negara - National Heart Institute, Kuala Lumpur
- Netherlands (7):
  - Universitair Medisch Centrum Groningen, Groningen
  - Zuyderland Medisch Centrum Heerlen, Heerlen
  - Maastricht Universitair Medisch Centrum (MUMC), Maastricht
  - St. Antonius Ziekenhuis, Nieuwegein
  - HagaZiekenhuis - Locatie Leyweg, The Hague
  - VieCuri Medisch Centrum voor Noord-Limburg - Locatie Venlo, Venlo
  - Isala Zwolle, Zwolle
- New Zealand (3):
  - Auckland City Hospital, Auckland
  - Waikato Hospital, Hamilton
  - Wellington Hospital, Newtown
- Norway (2):
  - Oslo Universitetssykehus-Ullevål Universitetssykehus, Oslo
  - Stavanger Universitetssjukehus - Helse Stavanger HF, Stavanger
- Poland (3):
  - Górnośląskie Centrum Medyczne im prof Leszka Gieca Śląskiego Uniwersytetu Medycznego w Katowicach, Katowice
  - Miedziowe Centrum Zdrowia, Lubin
  - Szpital Kliniczny Przemienienia Panskiego, Poznan
- Singapore (2):
  - National University Hospital, Singapore
  - Tan Tock Seng Hospital, Singapore
- Stredoslovensky Ustav Srdcovych a Cievnych Chorob a.s, Banská Bystrica, Slovakia
- South Korea (9):
  - Keimyung University Dongsan Medical Center, Daegu
  - Chonnam National University Hospital, Gwangju
  - Seoul National University Bundang Hospital, Seongnam-si
  - Severance Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul Saint Mary's Hospital, Seoul
  - Asan Medical Center, Seoul
  - Wonju Severance Christian Hospital, Wŏnju
- Spain (8):
  - Hospital Clínico Universitario Virgen de la Arrixaca, El Palmar, Murcia
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Tenerife
  - Hospital General Universitario de Alicante, Alicante
  - Hospital del Mar, Barcelona
  - Hospital Universitari Bellvitge, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Hospital Clinico Universitario de Salamanca, Salamanca
  - Hospital Universitario Marques de Valdecilla, Santander
- Sweden (5):
  - Gävle sjukhus, Gävle
  - Universitetssjukhuset Örebro, Örebro
  - Södersjukhuset, Stockholm
  - Karolinska University Hospital in Solna, Stockholm
  - Västmanlands Sjukhus, Västerås
- Switzerland (2):
  - Inselspital - Universitätsspital Bern, Bern
  - Cardiocentro Ticino, Lugano
- Siriraj Hospital, Bangkok, Thailand
- United Kingdom (8):
  - Cardiff and Vale University Health Board - University Hospital of Wales (UHW), Cardiff
  - Royal Infirmary of Edinburgh, Edinburgh
  - Royal Devon and Exeter NHS Foundation Trust, Exeter
  - Golden Jubilee National Hospital - NHS Trust, Glasgow
  - Royal Free Hospital, London
  - The James Cook University Hospital - South Tees Hospitals NHS, Middlesbrough
  - The Newcastle upon Tyne Hospitals NHS Foundation Trust - Freeman Hospital, Newcastle upon Tyne
  - Queen Alexandra Hospital, Portsmouth

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Campos CM, Mehran R, Capodanno D, Owen R, Windecker S, Varenne O, Stone GW, Valgimigli M, Hajjar LA, Kalil Filho R, Oldroyd K, Morice MC, Urban P, Abizaid A. Risk Burden of Cancer in Patients Treated With Abbreviated Dual Antiplatelet Therapy After PCI: Analysis of Multicenter Controlled High-Bleeding Risk Trials. Circ Cardiovasc Interv. 2024 Apr;17(4):e013000. doi: 10.1161/CIRCINTERVENTIONS.122.013000. Epub 2024 Apr 16. PMID 38626080
- [Derived] Toth GG, Kandzari DE, Kirtane AJ, Windecker S, Latib A, Kedhi E, Mehran R, Price MJ, Choi JW, Caputo R, Troquay R, Diderholm E, Singh S, Brar SS, Loussararian A, Chetcuti S, Tulli M, Stone GW, Lung TH, Mylotte D. Two-year results from Onyx ONE clear in patients with high bleeding risk on one-month DAPT with and without intracoronary imaging. Cardiovasc Revasc Med. 2024 Jan;58:60-67. doi: 10.1016/j.carrev.2023.07.016. Epub 2023 Jul 24. PMID 37550123
- [Derived] Windecker S, Latib A, Kedhi E, Kirtane AJ, Kandzari DE, Mehran R, Price MJ, Abizaid A, Simon DI, Worthley SG, Zaman A, Hudec M, Poliacikova P, Kahar Bin Abdul Ghapar A, Selvaraj K, Petrov I, Mylotte D, Pinar E, Moreno R, Fabbiocchi F, Pasupati S, Kim HS, Aminian A, Tie C, Wlodarczak A, Hur SH, Marx SO, Ali ZA, Parke M, Lung TH, Stone GW; Onyx ONE Investigators. Polymer-Based Versus Polymer-Free Stents in High Bleeding Risk Patients: Final 2-Year Results From Onyx ONE. JACC Cardiovasc Interv. 2022 Jun 13;15(11):1153-1163. doi: 10.1016/j.jcin.2022.04.010. PMID 35680195
- [Derived] Windecker S, Latib A, Kedhi E, Kirtane AJ, Kandzari DE, Mehran R, Price MJ, Abizaid A, Simon DI, Worthley SG, Zaman A, Hudec M, Poliacikova P, Abdul Ghapar AKB, Selvaraj K, Petrov I, Mylotte D, Pinar E, Moreno R, Fabbiocchi F, Pasupati S, Kim HS, Aminian A, Tie C, Wlodarczak A, Hur SH, Marx SO, Jankovic I, Brar S, Bousquette L, Liu M, Stone GW; ONYX ONE Investigators. Polymer-based or Polymer-free Stents in Patients at High Bleeding Risk. N Engl J Med. 2020 Mar 26;382(13):1208-1218. doi: 10.1056/NEJMoa1910021. Epub 2020 Feb 12. PMID 32050061
- [Derived] Kedhi E, Latib A, Abizaid A, Kandzari D, Kirtane AJ, Mehran R, Price MJ, Simon D, Worthley S, Zaman A, Brar S, Liu M, Stone GW, Windecker S. Rationale and design of the Onyx ONE global randomized trial: A randomized controlled trial of high-bleeding risk patients after stent placement with 1 month of dual antiplatelet therapy. Am Heart J. 2019 Aug;214:134-141. doi: 10.1016/j.ahj.2019.04.017. Epub 2019 May 6. PMID 31203158